CLINICAL TRIAL: NCT04013113
Title: A Randomized Controlled Trial of Efficacy and Safety of Hemoperfusion or Plasma Exchange Compared to Standard Medical Therapy in Patients With Acute on Chronic Liver Failure
Brief Title: Efficacy and Safety of Hemoperfusion or Plasma Exchange Compared to Standard Medical Therapy in Patients With Acute on Chronic Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-03
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Hemoperfusion; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Medical Treatment (Active Comparator): Group A will be given standard medical therapy only included as per requirement.nutritional therapy ( high calorie intake- 2400 Kcal/ day) Lactulose, bowel wash, albumin, terlipressin, antibiotics and anti-virals in hepatitis B reactivation will be continued and recorded.
  Interventions: Drug: Standard Medical Treatment
- Hemoadsorption plus standard medical therapy (Experimental)
  Interventions: Drug: Haemoperfusion; Drug: Standard Medical Treatment
- Plasma Exchange plus standard medical therapy (Experimental)
  Interventions: Drug: Standard Medical Treatment; Other: Plasma Exchange

INTERVENTIONS:
Drug: Haemoperfusion — Three sessions of Hemoperfusion, 1 plasma volume/session will be done to the selected patients.
  Hemoperfusion will be done through bile acids and ammonia filters to adsorb bile acids and ammonia respectively.
  Group specific fresh frozen plasma will be transfused to the patient through a peripheral vein catheter to prevent hypotension if required.
  Arms: Hemoadsorption plus standard medical therapy
Drug: Standard Medical Treatment — Standard medical therapy only included as per requirement.nutritional therapy ( high calorie intake- 2400 Kcal/ day) Lactulose, bowel wash, albumin, terlipressin, antibiotics and anti-virals in hepatitis B reactivation will be continued and recorded.
Other: Plasma Exchange — Fresh frozen plasma will be used as replacement fluid.TPE treatment shall be given on first day and continued on an a dailybasis/alternate day till the desired clinical or biochemical response is achieved.
  The procedures of TPE and hemoperfusion will be stopped if any major side effects occur (described below), the patient expires or the patient is transplanted within 30 days (whichever is earlier).
  Arms: Plasma Exchange plus standard medical therapy

SUMMARY:
The study is done with the aim of finding the association between the bilirubin and bile acids / DAMPS molecule with organ failures and sepsis in the patients with acute on chronic liver failure . in this study there are 2 parts in the first part people who satisfy the eligibility criteria will be recruited and blood samples will be taken and above mentioned molecules will be analyzed and association ,if any with occurrences of organ failures / new onset sepsis will be analyzed .

In the second part of the study the patients who meet the criteria will be randomized to either receive standard medical therapy or with either haemoperfusion or therapeutic plasma exchange with standard medical therapy . blood samples will be taken and stored, bile acids (primary and secondary bile acids, bilirubin and damps molecules will be analysed .the patients are followed for 90 days , then statistical analysis will be done to find the association with organ failures and new onset sepsis .

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ACLF as per APASL criteria will be included.
2. Age : 18-65 yrs.

Exclusion Criteria:

1. Patient with ischemic heart disease
2. Patient with chronic obstructive disease.
3. Patient with hepato cellular carcinoma.
4. Patient with extra hepatic malignancy.
5. Patient with chronic renal insufficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival in all the group | day 28

SECONDARY OUTCOMES:
Development of organ dysfunction in all the group | Day 7
Development of organ dysfunction in all the group | Day 15
Development of organ dysfunction in all the group | Day 28
New onset of sepsis in ll the groups | Day 7
New onset of sepsis in ll the groups | Day 15
New onset of sepsis in ll the groups | Day 28
Adverse Events in all the groups | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided